CLINICAL TRIAL: NCT01021475
Title: Does Visceral Manipulation Works in Treating Functional Dyspepsia? A Randomized Study
Brief Title: Does Visceral Manipulation Works in Treating Functional Dyspepsia?
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International College of Osteopathic Medicine (Other)
Responsible Party: Massimo Rossi DO BSc (student), ICOM
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VM-01
Record Dates: First submitted 2009-11-27; First posted 2009-11-30 (Estimated); Last update posted 2009-11-30 (Estimated); Status verified 2009-11

CONDITIONS: Functional Dyspepsia
Keywords: Functional Dyspepsia, Visceral Manipulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual drug FD therapy + Visceral Manipulation (Experimental)
  Interventions: Procedure: Visceral Manipulation
- Usual drug FD therapy (Active Comparator)
  Interventions: Drug: PPIs and/or Domperidone

INTERVENTIONS:
Procedure: Visceral Manipulation — Usual FD drug therapy (PPIs and/or Domperidone in base of symptom complain) for 4 weeks and 4 VM visits with weekly frequency with first VM visit at day 1 of drug therapy.
  Arms: Usual drug FD therapy + Visceral Manipulation
Drug: PPIs and/or Domperidone — Usual FD drug therapy (PPIs and/or Domperidone in base of symptom complain) for 4 weeks
  Arms: Usual drug FD therapy

SUMMARY:
The goal of this study is to determine if Visceral Manipulation (VM) is effective in treating Functional Dyspepsia in addition to drug therapy.

Null hypothesis is that VM does not influence FD symptoms.

DETAILED DESCRIPTION:
50 patients with Functional Dyspepsia (FD) diagnosed by General Practitioners are randomized in two therapy group: 1) drug only group and 2) drug + Visceral Manipulation group. Group 1 receive drug therapy for 4 weeks, Group 2 receive drug therapy for 4 weeks and 4 Visceral Manipulation visits with weekly frequency (visit 1 at day 1 of drug therapy). FD symptoms are recorded with VAS at baseline and after 1 and 4 weeks of therapy, and after 8 weeks (4 weeks after the finish of all therapies).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Functional Dyspepsia

Exclusion Criteria:

* Diabetes Mellitus
* Mental disturbance
* Thyroid gland dysfunction
* Intestinal, liver and biliary tract disease
* Concurrent medications that could interact with GI function
* Positive Helicobacter Pylori status

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
FD symptoms: Bothersome postprandial fullness / Early satiation / Epigastric pain / Epigastric burning | baseline, 1, 4 and 8 weeks after therapy start

CONTACTS AND LOCATIONS:
Overall Officials: Rossi Massimo, DO B.Sc (student), Principal Investigator — International College of Osteopathic Medicine
Locations (1):
- Ambulatori Comunali di Cavenago Brianza, Cavenago di Brianza, Milano, Italy